CLINICAL TRIAL: NCT02324543
Title: Phase 1/2 Study of Gemcitabine/Taxotere/Xeloda (GTX) in Combination With Cisplatin and Irinotecan in Subjects With Metastatic Pancreatic Cancer
Brief Title: Study of Gemcitabine/Taxotere/Xeloda (GTX) in Combination With Cisplatin and Irinotecan in Subjects With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Swim Across America (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J14161; J14161 (Other: Swim Across America Laboratory); IRB00053208 (Other: JHMIRB)
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Results first posted 2020-09-14 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
MeSH Terms: interventions — Gemcitabine; Docetaxel; Capecitabine; Cisplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Dose level 1 - Phase 1 (Experimental): * Gemcitabine - 400 mg/m^2
  * Taxotere - 20 mg/m^2
  * Xeloda - 500 mg/twice daily (BID)
  * Cisplatin - 15 mg/m^2
  * Irinotecan - 20 mg/m^2
  Interventions: Drug: Gemcitabine; Drug: Taxotere; Drug: Xeloda; Drug: Cisplatin; Drug: Irinotecan
- Dose Level 2 - Phase 1 (Experimental): * Gemcitabine - 400 mg/m^2
  * Taxotere - 20 mg/m^2
  * Xeloda - 500 mg/BID
  * Cisplatin - 15 mg/m^2
  * Irinotecan - 40 mg/m^2
  Interventions: Drug: Gemcitabine; Drug: Taxotere; Drug: Xeloda; Drug: Cisplatin; Drug: Irinotecan
- Dose Level 3 - Phase 1 (Experimental): * Gemcitabine - 400 mg/m^2
  * Taxotere - 20 mg/m^2
  * Xeloda - 500 mg/BID
  * Cisplatin - 15 mg/m^2
  * Irinotecan - 60 mg/m^2
  Interventions: Drug: Gemcitabine; Drug: Taxotere; Drug: Xeloda; Drug: Cisplatin; Drug: Irinotecan
- Dose Level 1a - Phase 1 (Experimental): * Gemcitabine - 500 mg/m^2
  * Taxotere - 20 mg/m^2
  * Xeloda - 500 mg/BID
  * Cisplatin - 20 mg/m^2
  * Irinotecan - 20 mg/m^2
  Interventions: Drug: Gemcitabine; Drug: Taxotere; Drug: Xeloda; Drug: Cisplatin; Drug: Irinotecan
- Dose level 1b - Phase 1 (Experimental): * Gemcitabine - 500 mg/m^2
  * Taxotere - 20 mg/m^2
  * Xeloda - 500 mg/BID
  * Cisplatin - 20 mg/m^2
  * Irinotecan - 40 mg/m^2
  Interventions: Drug: Gemcitabine; Drug: Taxotere; Drug: Xeloda; Drug: Cisplatin; Drug: Irinotecan
- Phase 2 (Experimental): * Gemcitabine - 500 mg/m^2
  * Taxotere - 20 mg/m^2
  * Xeloda - 500 mg/BID
  * Cisplatin - 20 mg/m^2
  * Irinotecan - 20 mg/m^2
  Interventions: Drug: Gemcitabine; Drug: Taxotere; Drug: Xeloda; Drug: Cisplatin; Drug: Irinotecan

INTERVENTIONS:
Drug: Gemcitabine — IV on days 4 and 11 of a 21 day cycle
  Other Names: Gemzar
Drug: Taxotere — IV on days 4 and 11 of a 21 day cycle
  Other Names: Docetaxel
Drug: Xeloda — Twice a day orally on days 1 through 14 of a 21 day cycle
  Other Names: Capecitabine
Drug: Cisplatin — IV on days 4 and 11 of a 21 day cycle
  Other Names: Platinol
Drug: Irinotecan — IV on days 4 and 11 of a 21 day cycle
  Other Names: Camptosar

SUMMARY:
This study will be looking at whether gemcitabine, taxotere, and xeloda (GTX) in combination with cisplatin and irinotecan is effective (anti-tumor activity) and safe in patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
The study is being done in 2 parts. The first part is the dose escalation (Phase I) part of the study where the dose of irinotecan is increased until the highest safe dose of irinotecan is defined that can be given with gemcitabine, taxotere, xeloda, and cisplatin.

After the safe dose of irinotecan in combination with gemcitabine, taxotere, xeloda, and cisplatin is defined, the second part of the study (Phase 2) will use these defined doses to look at how effective these drugs are against advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed untreated metastatic pancreatic adenocarcinoma.
2. Have measurable disease.
3. Male or non-pregnant and non-lactating female of age >18 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 . ECOG 0 indicates that the patient is fully active and able to carry on all pre-disease activities without restriction; and, ECOG 1 indicates that the patient is restricted in physically strenuous activity but is ambulatory and able to carry out work of a light or sedentary nature
5. Subjects must have adequate organ and marrow function.
6. Must use acceptable form of birth control prior to study and and for the duration of study.
7. Willing and able to comply with study procedures

Exclusion Criteria:

1. Patient who have had any prior chemotherapy within 5 years of enrollment.
2. Patient who have had radiotherapy for pancreatic cancer.
3. Age ≥ 76 years
4. Patient who is receiving or have received any other investigational agents within 28 days prior to Day 1 of treatment in this study.
5. Patient who has undergone major surgery, other than diagnostic surgery within 28 days prior to Day 1 of treatment in this study.
6. Patient who has known brain metastases.
7. Patient with history of hypersensitivity or allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine, taxotere, xeloda, cisplatin, or irinotecan.
8. Patient with uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
9. Patient who has serious medical risk factors involving any of the major organ systems.
10. Patient who has known history of infection with HIV, hepatitis B, or hepatitis C.
11. Pregnant or breast feeding.
12. Patient is unwilling or unable to comply with study procedures
13. Patient with clinically significant wound

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dung Le, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christenson ES, Lim SJ, Durham J, De Jesus-Acosta A, Bever K, Laheru D, Ryan A, Agarwal P, Scharpf RB, Le DT, Wang H. Cell-free DNA Predicts Prolonged Response to Multi-agent Chemotherapy in Pancreatic Ductal Adenocarcinoma. Cancer Res Commun. 2022 Nov 11;2(11):1418-1425. doi: 10.1158/2767-9764.CRC-22-0343. eCollection 2022 Nov. PMID 36970054

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1- Phase 1: Gemcitabine: 400 mg/m^2 IV on days 4 and 11 of a 21 day cycle
  Taxotere: 20 mg/m^2 IV on days 4 and 11 of a 21 day cycle
  Xeloda: 500 mg/BID twice a day orally on days 1-14 of a 21 day cycle
  Cisplatin: 15 mg/m^2 IV on days 4 and 11 of a 21 day cycle
  Irinotecan: 20 mg/m^2 IV on days 4 and 11 of a 21 day cycle
- Dose Level 1a - Phase 1; Phase 2: Gemcitabine: 500 mg/m^2 IV on days 4 and 11 of a 21 day cycle
  Taxotere: 20 mg/m^2 IV on days 4 and 11 of a 21 day cycle
  Xeloda: 500 mg/BID twice a day orally on days 1-14 of a 21 day cycle
  Cisplatin: 20 mg/m^2 IV on Days 4 and 11 of a 21 day cycle
  Irinotecan: 20 mg/m^2 IV on days 4 and 11 of a 21 day cycle
- Dose Level 1b - Phase 1: Gemcitabine - 500 mg/m^2 IV on days 4 and 11 of a 21 day cycle
  Taxotere - 20 mg/m^2 IV on days 4 and 11 of a 21 day cycle
  Xeloda - 500 mg/BID twice a day orally on days 1-14 of a 21 day cycle
  Cisplatin - 20 mg/m^2 IV on days 4 and 11 of a 21 day cycle
  Irinotecan - 40 mg/m^2 IV on days 4 and 11 of a 21 day cycle
- Dose Level 2 - Phase 1: Gemcitabine - 400 mg/m^2 IV on days 4 and 11 of a 21 day cycle
  Taxotere - 20 mg/m^2 IV on days 4 and 11 of a 21 day cycle
  Xeloda - 500 mg/BID twice a day orally on days 1-14 of a 21 day cycle
  Cisplatin -15 mg/m^2 IV on days 4 and 11 of a 21 day cycle
  Irinotecan - 40 mg/m^2 IV on days 4 and 11 of a 21 day cycle
- Dose Level 3 - Phase 1: Gemcitabine - 400 mg/m^2 IV on days 4 and 11 of a 21 day cycle
  Taxotere - 20 mg/m^2 IV on days 4 and 11 of a 21 day cycle
  Xeloda - 500 mg/BID twice a day orally on days 1-14 of a 21 day cycle
  Cisplatin - 15 mg/m^2 IV on days 4 and 11 of a 21 day cycle
  Irinotecan - 60 mg/m^2 IV on days 4 and 11 of a 21 day cycle
Period: Overall Study
Arm/Group | Dose Level 1- Phase 1 | Dose Level 1a - Phase 1 | Dose Level 1b - Phase 1 | Dose Level 2 - Phase 1 | Dose Level 3 - Phase 1 | Phase 2
Started | 6 | 6 | 3 | 4 | 4 | 24
Completed | 6 | 6 | 3 | 4 | 4 | 24
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 1 - Phase 1: Gemcitabine: 400 mg/m^2 IV on days 4 and 11 of a 21 day cycle
  Taxotere: 20 mg/m^2 IV on days 4 and 11 of a 21 day cycle
  Xeloda: 500 mg/BID twice a day orally on days 1-14 of a 21 day cycle
  Cisplatin: 15 mg/m^2 IV on days 4 and 11 of a 21 day cycle
  Irinotecan: 20 mg/m^2 IV on days 4 and 11 of a 21 day cycle
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 - Phase 1 | Dose Level 1a - Phase 1 | Dose Level 1b - Phase 1 | Dose Level 2 - Phase 1 | Dose Level 3 - Phase 1 | Phase 2 | Total
Number analyzed (Participants) | 6 | 6 | 3 | 4 | 4 | 24 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 2 | 4 | 2 | 13 | 26
  >=65 years | 3 | 4 | 1 | 0 | 2 | 11 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 1 | 1 | 3 | 8 | 20
  Male | 2 | 3 | 2 | 3 | 1 | 16 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 6 | 3 | 4 | 4 | 23 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 1 | 2 | 5
  White | 6 | 4 | 3 | 2 | 3 | 22 | 40
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Gemcitabine
Description: Dose escalation (phase I portion of the trial only) to determine the MTD in mg/m^2.
Time Frame: 28 days
Measure: Number; unit: mg/m^2
Groups:
- Phase 1: Gemcitabine: 500 mg/m^2 IV on days 4 and 11 of a 21 day cycle
  Taxotere: 20 mg/m^2 IV on days 4 and 11 of a 21 day cycle
  Xeloda: 500 mg/BID twice a day orally on days 1-14 of a 21 day cycle
  Cisplatin: 20 mg/m^2 IV on Days 4 and 11 of a 21 day cycle
  Irinotecan: 20 mg/m^2 IV on days 4 and 11 of a 21 day cycle
Arm/Group | Phase 1
Number analyzed (Participants) | 23
mg/m^2 | 500

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Docetaxel
Description: Dose escalation (phase I portion of the trial only) to determine the MTD in mg/m^2.
Time Frame: 28 days
Measure: Number; unit: mg/m^2
Arm/Group | Phase 1
Number analyzed (Participants) | 23
mg/m^2 | 20

3. Primary Outcome: Maximum Tolerated Dose (MTD) of Capecitabine
Description: Dose escalation (phase I portion of the trial only) to determine the MTD in mg for twice daily (BID) use.
Time Frame: 28 days
Measure: Number; unit: mg
Arm/Group | Phase 1
Number analyzed (Participants) | 23
mg | 500

4. Primary Outcome: Maximum Tolerated Dose (MTD) of Cisplatin
Description: Dose escalation (phase I portion of the trial only) to determine the MTD in mg/m^2.
Time Frame: 28 days
Measure: Number; unit: mg/m^2
Arm/Group | Phase 1
Number analyzed (Participants) | 23
mg/m^2 | 20

5. Primary Outcome: Maximum Tolerated Dose (MTD) of Irinotecan
Description: Dose escalation (phase I portion of the trial only) to determine the MTD in mg/m^2.
Time Frame: 28 days
Measure: Number; unit: mg/m^2
Arm/Group | Phase 1
Number analyzed (Participants) | 23
mg/m^2 | 20

6. Primary Outcome: Overall Survival (OS) Rate at 9 Months
Description: OS will be measured as the percentage of subjects alive at 9 months. (OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis). Estimation based on the Kaplan-Meier curve. (Phase 2 data only)
Time Frame: 9 months
Population: This measure was only assessed for Phase 2. Per protocol, the 6 subjects treated at the MTD (DL1a) during dose escalation (Phase 1) were counted toward the total sample size of 30 subjects for the Phase 2 outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2
Number analyzed (Participants) | 30
percentage of participants | 57 [41 to 77]

7. Secondary Outcome: Response Rate (RR) Using RECIST 1.1 Criteria
Description: RR is defined as the percentage of participants achieving a complete response (CR) or partial response (PR) based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) at any time during the study. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Time Frame: 43 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2
Number analyzed (Participants) | 30
percentage of participants | 57 [37 to 75]

8. Secondary Outcome: Disease Control Rate (DCR) Using RECIST 1.1 Criteria
Description: DCR is defined as the percentage of participants achieving a complete response (CR) or partial response (PR) and stable disease (SD) based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) at any time during the study. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Time Frame: 43 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2
Number analyzed (Participants) | 30
percentage of participants | 87 [69 to 96]

9. Secondary Outcome: Progression-free Survival (PFS) Using RECIST 1.1 Criteria
Description: PFS is defined as the number of months from the date of first dose to disease progression (progressive disease [PD] or relapse from complete response [CR] as assessed using RECIST 1.1 criteria) or death due to any cause. Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on the Kaplan-Meier curve.
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2
Number analyzed (Participants) | 30
Months | 8.34 [6.34 to NA] — Upper bound confidence interval was not reached.

10. Secondary Outcome: Overall Survival (OS)
Description: OS will be measured (in months) from date of first dose until death or end of follow-up (OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis). Estimation based on the Kaplan-Meier curve.
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2
Number analyzed (Participants) | 30
Months | 11.02 [8.54 to 21.09]

ADVERSE EVENTS:
Time Frame: All adverse events will be collected from the first dose up to 30 days after last dose.
Arm/Group | Dose Level 1 - Phase 1 | Dose Level 1a - Phase 1 | Dose Level 1b - Phase 1 | Dose Level 2 - Phase 1 | Dose Level 3 - Phase 1 | Phase 2
All-Cause Mortality (participants affected / at risk) | 2/6 | 1/6 | 0/3 | 0/4 | 0/4 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 1/3 | 2/4 | 1/4 | 2/24
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 3/3 | 4/4 | 4/4 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 - Phase 1 (N=6) | Dose Level 1a - Phase 1 (N=6) | Dose Level 1b - Phase 1 (N=3) | Dose Level 2 - Phase 1 (N=4) | Dose Level 3 - Phase 1 (N=4) | Phase 2 (N=24)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 - Phase 1 (N=6) | Dose Level 1a - Phase 1 (N=6) | Dose Level 1b - Phase 1 (N=3) | Dose Level 2 - Phase 1 (N=4) | Dose Level 3 - Phase 1 (N=4) | Phase 2 (N=24)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 4 (4) | 2 (2) | 1 (1) | 2 (2) | 14 (14)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 6 (6)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 3 (3) | 3 (3) | 3 (3) | 4 (4) | 17 (17)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 6 (6)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 12 (12)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4) | 1 (1) | 2 (2) | 2 (2) | 9 (9)
Edema (General disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 4 (4) — and administration site conditions
Fatigue (General disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 16 (16) — and administration site conditions
Fever (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (5) — and administration site conditions
Sweating (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — and administration site conditions
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Creatinine, increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (16)
Lymphocyte count decreased (Investigations) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 9 (9)
Neutrophil count decreased (Investigations) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 3 (3) | 15 (15)
Platelet count decreased (Investigations) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 9 (9)
Weight Loss (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
White blood count decreased (Investigations) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 12 (12)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 6 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 3 (3) | 2 (2) | 3 (3) | 15 (15)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 17 (17)
Neuropathy (Nervous system disorders) | 3 (3) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 15 (15)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 6 (6)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 12 (12)
Dry Skin (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 7 (7)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cold Intolerance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — and administration site conditions
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Early satiety (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nail Loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth sensitivity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight gain (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT02324543/Prot_SAP_000.pdf